CLINICAL TRIAL: NCT05208879
Title: Characterization of the Density of Macular Pigment in Patients With Primary Intestinal Hypocholesterolemia and Its Relation to Their Carotenoid and Anti-oxidant Status.
Brief Title: CArotenoid in hypoChOlesterolemia
Acronym: CaCo
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0720
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Primary Intestinal Hypocholesterolemia; Abetalipoproteinemia; Chylomicron Retention Disease
Keywords: Abetalipoproteinemia,; Chylomicron Retention Disease; Hypocholesterolemia; Macula Pigment; Retinitis Pigmentosa; Carotenoids
MeSH Terms: conditions — Abetalipoproteinemia; Chylomicron retention disease; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group.: Patients with genetically proven familial hypocholesterolemia, who will accept to participate in this study and have been treated for this pathology since 1990 in the Department of Gastroenterology and Paediatric Nutrition (Pr Peretti) and continue their follow-up into adulthood at the GHE (Groupement Hospitalier Est) in Lyon in the endocrinology-nutrition service (Pr Moulin).
  They may be girl/woman or boy/man over 6 years of age and over 12 kg at the time of inclusion (age required for cooperation on macular pigment measurement), agreeing to participate in the study with clear and informed consent. These patients are covered by social security.
  Interventions: Biological: Characterization of carotenoid status and plasma levels of oxidative stress markers in patients (case group only)
- Control group.: The control group consists of children over 6 years old or adult patients, followed routinely in the ophthalmology department of the Edouard Herriot Hospital, Lyon (Pr Kodjikian) not suffering from genetic hypocholesterolemia and requiring a fundus examination as part of the usual follow-up of their ocular pathology, if this pathology does not interfere with the macular pigment density. An additional measurement of the macular pigment density will be made during this examination. The control group is only needed for the macular pigment analysis. No control group is considered for the characterization of plasma lutein and zeaxanthin deficiency and for the analysis of oxidative stress, so there will be no additional blood sampling for control patients.
  Interventions: Other: Characterization, evaluation and comparison of macular pigment density

INTERVENTIONS:
Biological: Characterization of carotenoid status and plasma levels of oxidative stress markers in patients (case group only) — Carotenoid status will be determined by measuring plasma and erythrocyte concentrations of lutein and zeaxanthin obtained during an annual blood draw. These molecules will be analyzed by high performance liquid chromatography.
  The oxidative stress markers will be measured, in the blood sample already collected, thanks to specific assay kits: Erythrocyte reduced glutathione, Superoxide dismutase (SOD), Glutathione peroxidase (GPx), Plasma and erythrocyte malondialdehyde, Plasma vitamin C, Plasma oxidized cholesterol, F2-isoprostanes.
  This study does not result in any change in patient management, but requires the collection of an additional volume of blood (14 ml of study-specific blood) during the annual blood draw performed as part of routine patient follow-up.
  Groups: Case group.
Other: Characterization, evaluation and comparison of macular pigment density — The macular pigment optical density (OD) will be determined by an additional photograph during the fundus usually performed for annual follow-up through two-wavelength autofluorescence imaging. Indeed, the measurement of the optical density consists of an additional post-examination analysis of additional retinal images obtained during the fundus performed for the patients' ophthalmologic follow-up.
  Groups: Control group.

SUMMARY:
Hypobetalipoproteinemias (HBL) represent a heterogeneous group of disorders characterized by reduced plasma levels of plasmatic lipids (mainly triglycerides, total cholesterol (TC), LDL-cholesterol (LDL-C), and apolipoprotein B (apoB)) below the 5th percentile of the general population adjusted for age, gender. HBL may be attributed to inherited disorders caused by mutations in several known genes. Intestinal recessive HBL includes abetalipoproteinemia (ABL) (OMIM 200100) and Chylomicron Retention Disease (CMRD) (OMIM 246700) - also called Anderson's disease. Those two recessives form of HBL are the ones considered in this study. ABL is due to mutations in the Microsomal Triglyceride Transfer Protein (MTTP) gene which is required for the assembly and secretion of apoB-containing lipoproteins: Low-Density Lipoprotein (LDL) and chylomicrons (CM) in both liver and intestine. Similarly, CMRD is due to mutations in the Sar1b gene encoding the Sar1b protein involved in the control of the intracellular trafficking of CMs in COPII-coated vesicles. Due to a defect in Apolipoprotein B-containing lipoproteins these diseases are characterized by dietary lipids and fat-soluble vitamins (A, D, E, K) malabsorption inducing digestive and growth disorders from birth. In parallel, neurological manifestations may appear, mainly as a consequence of vitamin E and A deficiencies.

Ophthalmological disorders are inconstant, with many patients being asymptomatic until adulthood. Loss of night or color vision are the first symptoms associated with retinal degeneration. Without treatment with high doses of vitamins, retinal degeneration can lead to blindness. The exact biological mechanism still remains unknown. Indeed, cases described in the scientific literature demonstrate that early treatment with high doses of vitamin E and A can stop or prevent neurological complications in the vast majority of patients; however, ophthalmic complications have a more versatile response.

Thus, despite early vitamin supplementation, several cases of adolescent or adult patients with vision impairment in the form of retinitis pigmentosa have been reported. This so-called secondary retinitis pigmentosa is characterized by a progressive loss of photoreceptors and a dysfunction of the pigmentary epithelium resulting in a progressive and gradual loss of vision, usually leading to blindness. Interestingly, primary (i.e., genetic) retinitis pigmentosa are characterized by "macula lutea" atrophy composed of two lipophilic molecules from the carotenoid xanthophyll family lutein and zeaxanthin, also known as macular pigments. Moreover, preliminary data seem to show that the patients considered for this study, present decreased plasmatic carotene concentrations as well as plasmatic vitamin E concentrations largely lower than the threshold of normality.

Thus, even if early treatment seems to prevent major ophthalmic complications, it does not provide total ophthalmic protection, which suggests the involvement of other factors among which carotenoids could occupy a prominent place given their essential role in maintaining the integrity of the macula.

ELIGIBILITY:
Inclusion Criteria:

* Genetically proven family hypocholesterolemia patients,
* Patients systematically monitored in the Gastroenterology and Paediatric Nutrition department of the Women's Hospital Mother Child of Lyon or in the adult endocrinology department of the GHE (Louis Pradel Hospital),
* Girl/woman or boy/man over 6 years and over 12 kg at the time of inclusion (age required for cooperation on macular pigment measurement),
* No objection from the patient or their parents/legal tutors in the case of a minor patient,
* Patient covered by social security.

Exclusion Criteria:

* Allergy to local anesthetics (especially xylocaine)
* Mydriatic allergy
* Person participating in another research with an exclusion period still in progress at pre-inclusion
* Person subject to a safeguard measure.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study relates to adults or children over 6 years of age (cooperation necessary to perform the fundus) with primary intestinal hypocholesterolemia.
  The control population comprising major control patients under the age of 50 (limit the risk of age-related macular degeneration - AMD) or under age over 6 (cooperation necessary to perform OF) routinely monitored in the service of ophthalmology requiring a fundus examination as part of their usual follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
The principal outcome measure is the macular pigment optical density (OD) | The optical density measurement will be performed, in addition to the usual patient follow-up tests, during a single visit to the ophthalmology department on a date chosen by the patient.
  The macular pigment optical density (OD) will be determined by an additional photograph during the fundus usually performed for annual follow-up through two-wavelength autofluorescence imaging. This imaging method provides a profile of autofluorescence distribution calculated using a gray intensity scale in the center of the macula and along the horizontal and vertical meridians. The optical density of the macular pigment is then expressed as the logarithm of the ratio of the peri-oval/foveal excitation spectra symbolized by the acronym "DU" ("Density Unit"). Indeed, in autofluorescence, the lipofuscin chromophores are generally excited with two wavelengths: a first one which is located in the blue spectral region where the absorption band of the lipofuscin overlaps that of the macular pigments, and a second one which is always located in the absorption region of the lipofuscin but outside the absorption range of the macular pigments. Thus, excitation by the first (green) light causes

CONTACTS AND LOCATIONS:
Overall Officials: Peretti Noël, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Fédération d'endocrinologie, maladies métaboliques, diabète et nutrition Hôpital cardiovasculaire et pneumologique Louis Pradel, Bron, Bron
  - UF nutrition pédiatrique, Service hépatologie, gastroentérologie et nutrition pédiatrique Hôpital Femme Mère Enfant de Lyon (GHE-HFME), Bron, Bron
  - UF nutrition pédiatrique, Service hépatologie, gastroentérologie et nutrition pédiatrique Hôpital Femme Mère Enfant de Lyon (GHE-HFME), Bron